CLINICAL TRIAL: NCT04250688
Title: Effect of a Robotic Exoskeleton With Functional Electrical Stimulation on Neural Recovery in Individuals With Acute Spinal Cord Injury
Brief Title: Robotic Exoskeleton With Functional Electrical Stimulation in Acute Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STU00202078
Record Dates: First submitted 2020-01-28; First posted 2020-01-31 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Spinal Cord Injuries
Keywords: exoskeleton; ambulation; robotics; Functional electrical stimulation; acute spinal cord injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Esko Bionics Suit + Functional Electrical Stimulation (Experimental)
  Interventions: Device: Ekso Training with FES
- Control (No Intervention)

INTERVENTIONS:
Device: Ekso Training with FES
  Arms: Esko Bionics Suit + Functional Electrical Stimulation

SUMMARY:
The purpose of this study is to examine the effectiveness of mobility training using the Ekso robotic exoskeleton with functional electrical stimulation (FES) in persons affected by spinal cord injury; designated AIS classification A, B, C, or D. Traditionally, a person with an American Spinal Injury Association Impairment Scale (AIS) "A" injury, walking training is not performed. Even with AIS B, C and D injuries, although walking training may be appropriate, a person may not walk as much as needed to see an improvement due to environmental and staff limitations. The Ekso is a tool to give walking training to patients. The investigators aim to see if utilizing these technologies will affect recovery; specifically in sensation and muscle activity below the level of the injury as well as the ability to walk.

The Ekso is a wearable, battery- operated exoskeleton that assists with walking. The Ekso has motors at the hip and knee joints to provide assistance that may be needed with walking. All motion is initiated either through body weight shifts or the use of an external controller. The Ekso robotic exoskeleton has been approved by the Food and Drug Administration as a powered exercise device for rehabilitative purposes such as this study. Currently, the Ekso is approved for people with spinal cord injuries from T4-L5 given bilateral arm strength of 4/5. With injuries from C7-T3, individuals must have AIS classification of D with bilateral arm strength of 4/5. For this study, it is possible that Ekso GT will be used outside of the current FDA approval if the injury level is C7-T3 and the person is classified as an AIS A, B or C injury level. Functional electrical stimulation (FES) will be used in conjunction with the robotic exoskeleton. FES involves using surface electrodes placed on the skin like a sticker over key leg muscles that will be stimulated in the normal walking pattern as a person walks in the device.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effectiveness of mobility training using the Ekso robotic exoskeleton with functional electrical stimulation (FES) on neural recovery in individuals with acute spinal cord injury with American Spinal Injury Association Impairment Scale (AIS) neurologic classification A, B, C or D.

Specifically, individuals with acute SCI in the inpatient rehabilitation setting improve their AIS score after mobility training with the Ekso-FES compared to a control intervention period?

In addition, the investigators will analyze the influence of training performed early or later in acute rehabilitation phase on muscle properties, neural recovery and function.

This is an investigational clinical study trialing the efficacy of the Ekso device with FES in the acute SCI population. Participants with a diagnosis of spinal cord injury classified as AIS A, B, C or D will be included. Up to ten participants will be recruited to participate in this study. This number was arbitrarily chosen as this is an investigational study and there is no previous data on the Ekso device to specifically select subject number based on a power analysis. Participants will be recruited from inpatient units at The Shirley Ryan AbilityLab. Following screening, all subjects will be required to receive medical clearance from their attending inpatient physician.

Subjects will be randomized to which order they receive the Ekso intervention (A) and control (B) period (A then B or B then A). The device will be used in the lab and there will be no charge associated with use of the Ekso device.

All participants involved in the investigational study/training will be screened according to general inclusion/exclusion criteria after obtaining informed consent and before using the Ekso device.

Screening will include:

* Range of Motion (ROM): Range of motion of the joints of the upper and lower extremities will be measured using a goniometer
* Muscle strength testing: upper and lower extremity manual muscle testing to determine qualification for study inclusion.
* Modified Ashworth Scale (MAS): The Modified Ashworth Scale is a 6 point ordinal scale used to grade the amount of hypertonicity in individuals with neurological diagnoses. A score of 0 on the scale indicates no increase in tone while a score of 4 indicates rigidity. Tone is scored by passively moving the individual's limb and assessing the amount of resistance to movement felt by the examiner.
* Upper and lower leg length and hip measurements will be performed to determine safe fit in the exoskeleton device.

ELIGIBILITY:
Inclusion Criteria:

* Medical clearance from attending inpatient physician
* Have an upper motor neuron spinal cord injury classified as ASIA A, B or C or D between C7-T11Subacute injury <6 months at completion of study
* Be between 18-70 years of age.
* Be able to physically fit into the exoskeletal device.
* Be able to tolerate upright standing for a minimum of 30 minutes.
* Have joint range of motion within normal functional limits for ambulation.
* Have sufficient upper body strength to balance themself using the walker while wearing the exoskeleton.

Exclusion Criteria:

* Cervical level spinal cord injury above C6 or T12 and below
* Weight above 220 pounds
* Femur length above 47 cm or below 36 cm
* Joint contractures at the hip, knee, or ankle that limit normal range of motion (ROM) during ambulation;
* Cognitive and/or communication disability (e.g. due to brain injury);
* History of significant problems with skin break down or current skin break down that would prevent wearing the device;
* Any medical issue that precludes full weight bearing and ambulation (e.g. orthopedic injuries, pain, severe spasticity);
* History of severe osteoporosis or high risk of fractures. Medical clearance will be obtained for patients who are at risk of osteoporosis or fractures;
* Pregnancy;
* Inability to sign consent form indicating insufficient hand dexterity to utilize an assistive device.
* Cardiac Pacemaker;
* Metal implants in the areas of stimulation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in 6 Minute Walk Test from baseline in distance, rate of perceived exhaustion (RPE) | [Time Frame: Testing Day 1 - 3 and follow up testing Week 3 and Week 6.]
  The goal is to cover as much ground as possible over 6 minutes, the distance is measured with a measuring wheel. The minimum score is zero feet walked, there is no maximum score and the participant will be scored by how far they can walk in 6 minutes. The farther they walk, the better the score. The instructions are "Walk continuously if possible, but do not be concerned if you need to slow down or stop to rest." At the end of 6 minutes the participant is asked to rate their exertion level on a Borg Scale of 6 - 20 points.
Change in 10 meter walk test from baseline in gait speed | Time Frame: Testing Day 1 - 3 and follow up testing Week 3 and Week 6
  Measure the time in second for and individual to walk 10 meters. The test is performed using a "flying start," patient walks 10 meters (33 ft) and the time is measured when the leading foot crosses the start line and the finish line. The instructions are: " Please walk this distance as fast as you safely can when I say go."

SECONDARY OUTCOMES:
Magnetic resonance imaging lower extremity muscle volume | Time Frame: Testing Day 1 - 3 and follow up testing Week 3 and Week 6
  Manual segmentation of lower extremity musculature, for the purpose of muscle architectural quantification. Muscle's percent change was being compared
Magnetic resonance imaging lower extremity fat infiltration | Time Frame: Testing Day 1 - 3 and follow up testing Week 3 and Week 6
  Manual segmentation of lower extremity fat infiltration, for the purpose of muscle architectural quantification. Muscle's percent change was being compared

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab

IPD SHARING:
Plan to Share IPD: Undecided